CLINICAL TRIAL: NCT03898609
Title: Effect of Low-Fat Compared to Low-Carbohydrate Diet on Fasting Lipids and Metabolic Profile in Subjects With Multifactorial Chylomicronemia: A Randomized Crossover Study
Brief Title: Effect of Low-Fat Compared to Low-Carbohydrate Diet in Subjects With Multifactorial Chylomicronemia
Acronym: MCMdiet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Sophie Bernard, Director of the Lipids, Nutrition and Cardiovascular Prevention Clinic of the Montreal Clinical Research Institute (IRCM), Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019-957
Record Dates: First submitted 2019-03-25; First posted 2019-04-02 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Multifactorial Chylomicronemia (MCM)
MeSH Terms: interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-fat diet (Experimental): 20% fat 20% protein 60% carbohydrate
  Interventions: Other: Dietary intervention
- Low-carbohydrate diet (Experimental): 45% fat 20% protein 35% carbohydrate
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — 3 weeks

SUMMARY:
Introduction. The multifactorial chylomicronemia ((MCM), also known as type V hyperlipoproteinaemia or mixed hyperlipidaemia) is an oligogenic or polygenic disorder that is associated with a reduction in lipoprotein lipase activity which leads to chylomicronemia. In this disease, very high concentrations of serum triglycerides (≥10 mmol/l (≥880 mg/dL)) can be observed in the fasting state due to the accumulation of both VLDL-C and chylomicron. In patients with MCM, chylomicronemia typically occur in adulthood and is exacerbated by the presence of secondary factors such as a diet rich in dietary fats and simple sugars, obesity, alcohol intake and uncontrolled diabetes. It has been estimated that chylomicronemia can be found in 1:600 adults. However, it is likely that the prevalence of MCM may increase in the future due to the increasing prevalence of obesity, metabolic syndrome and type 2 diabetes. This condition increases the risk of acute pancreatitis, which can be recurrent and potentially fatal. Indeed, the risk of acute pancreatitis is 10-20% for TG levels > 22.58 mmol/L (>2000 mg/dL). Furthermore, because MCM patients often present with other lipid disturbances as well as a worse metabolic profile, these patients are at increased risk of cardiovascular disease (CVD). Fortunately, MCM patients generally respond well to modifications in lifestyle, to treatment of secondary factors and to triglycerides lowering therapies such as fibrates. However, it is still unknown which kind of diet has the greatest effect on triglycerides level and on the metabolic profile in MCM patients.

The nutritional recommendations can be very different according to the nature of the patient's population to be treated. In order to reduce and manage triglycerides level in the general population, the American Heart Association guidelines recommend reduction of simple carbohydrates intake.

On the other hand, the nutritional intervention strategy is quite different for subjects affected by familial chylomicronemia syndrome (FCS), for which the treatment focuses on restriction of dietary fat. FCS is a very rare autosomal recessive disease that leads to a drastic reduction of chylomicrons clearance leading to chylomicronaemia. Therefore, a very strict lipid-controlled diet low in long-chain fatty acid (10-30g/day or 10%-15% of total energy intake) is required in order to lower chylomicron formation.

MCM is a complex condition in which both an increased VLDL formation by the liver and a decreased chylomicrons and VLDL clearance are present. Furthermore, triglycerides values are fluctuating from day to day but generally remain very high. Therefore, the best dietary approach for these patients remains to be elucidated.

Primary Objective. The primary objective of this study is to compare the effects of low-fat vs low-carbohydrate diets on fasting serum triglyceride concentrations.

Secondary Objectives.

1. To compare the effects of low-fat vs low-carbohydrate diets on other fasting cardiometabolic parameters: measured LDL-C, total cholesterol, HDL-C, glucose, insulin, HOMA-IR, apoB, non-HDL-C, hs-CRP, PCSK9 and free fatty acids (FFA).
2. To compare the effects of low-fat vs low-carbohydrate diets on SBP, DBP and waist circumference.
3. To compare the effects of low-fat vs low-carbohydrate diets on lipoprotein subfractions (fasting).
4. To compare the effects of low-fat vs low-carbohydrate meals on postprandial triglycerides, insulin, glucose, FFA and PCSK9 after a standardized test meal.
5. To assess the patients' appreciation, compliance and tolerability for each experimental diet (feedback questionnaire).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 years.
2. Fasting triglycerides values ≥ 10 mmol/L (≥ 880 mg/dL) at least once, with or without medication.
3. Fasting triglycerides values ≥ 6.0 mmol/L at screening.

Exclusion Criteria:

1. A diagnosis of familial chylomicronemia syndrome, familial hypercholesterolemia or type III hyperlipidemia.
2. An episode of accute pancreatitis in the 6 months prior the screening.
3. Recent changes (in the last 3 months) in medication or supplement known to affect glucose metabolism such as steroid or oral contraceptive.
4. Recent changes (in the last 4 weeks) in lipid-lowering medication such as fibrates and statins.
5. Any condition known to affect lipid or glucose metabolism such as uncontrolled hypothyroidism or Cushing's syndrome.
6. Major surgery in the 3 months preceding the study.
7. Significant weight change (±10 %) within 3 months prior to beginning the study.
8. Inability to reduce alcohol use (0-2 units per week).
9. The necessity or the wish to follow a specific diet.
10. BMI ≥ 40 kg/m2.
11. Breastfeeding woman.
12. Pregnancy or the wish to become pregnant.
13. Consumption of dietary supplements such as omega-3, psyllium or phytosterols.
14. Any serious health condition associated with a life expectancy of ≤ 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change of triglycerides from baseline | 3 weeks
  Fasting serum triglyceride concentrations (mmol/L)

SECONDARY OUTCOMES:
Change of measured LDL-C from baseline | 3 weeks
  Fasting measured LDL-C concentrations (mmol/L)
Change of total cholesterol from baseline | 3 weeks
  Fasting total cholesterol concentrations (mmol/L)
Change of HDL-C from baseline | 3 weeks
  Fasting HDL-C concentrations (mmol/L)
Change of glucose from baseline | 3 weeks
  Fasting glucose concentrations (mmol/L)
Change of insulin from baseline | 3 weeks
  Fasting insulin concentrations (pmol/L)
Change of apolipoprotein B from baseline | 3 weeks
  Fasting apolipoprotein B concentrations (g/L)
Change of hs-CRP from baseline | 3 weeks
  Fasting hs-CRP concentrations (mg/L)
Change of PCSK9 from baseline | 3 weeks
  Fasting PCSK9 concentrations (ng/mL)
Change of free fatty acids from baseline | 3 weeks
  Fasting free fatty acids concentrations (mEq/L)
Change of systolic blood pressure from baseline | 3 weeks
  Measurement of systolic blood pressure (mmHg)
Change of diastolic blood pressure from baseline | 3 weeks
  Measurement of diastolic blood pressure (mmHg)
Change of waist circumference from baseline | 3 weeks
  Measurement of waist circumference (cm)
Change in the composition of lipoprotein fractions from baseline | 3 weeks
  Ultracentrifugation and lipoprotein electrophoresis
Postprandial triglycerides | One day
  After a standardized test meal (1h, 2h, 4h and 6h) (mmol/L)
Postprandial insulin | One day
  After a standardized test meal (1h, 2h, 4h and 6h) (pmol/L)
Postprandial glucose | One day
  After a standardized test meal (1h, 2h, 4h and 6h) (mmol/L)
Postprandial free fatty acids | One day
  After a standardized test meal (1h, 2h, 4h and 6h) (mEq/L)
Postprandial PCSK9 | One day
  After a standardized test meal (1h, 2h, 4h and 6h) (ng/mL)
Questionnaire of appreciation, compliance and tolerability | 3 weeks
  The patients' appreciation, compliance and tolerability for each experimental diet will be collected in a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Bernard, MD, PhD, Principal Investigator — Institut de Recherches Cliniques de Montreal (IRCM)
Locations (1):
- Institut de recherches cliniques de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No